CLINICAL TRIAL: NCT00528788
Title: Effect of Doxercalciferol on Endothelial Cell Function in End Stage Renal Disease
Brief Title: How Vitamin D Analogues Affect Endothelial Cells in Patients on Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001559
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2012-08

CONDITIONS: Hyperparathyroidism, Secondary; Kidney Failure, Chronic
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre and post doxicalciferol (Experimental): ESRD: all patients with secondary hyperparathyroidism who are vitamin D naive will receive doxercalciferol 2 mcg or 4 mcg 3 times per week fopr 30 days (1 month). Blood work and vascular laboratory studies will be performed pre and post treatment.
  Interventions: Drug: doxercalciferol

INTERVENTIONS:
Drug: doxercalciferol

SUMMARY:
Patients with chronic kidney disease and end stage renal disease have greater cardiovascular risk than the general population. Vitamin D analogues have been shown in observational studies to have mortality benefit for these patients. This study is designed to investigate doxercalciferol's effect on the vasculature (i.e. endothelial cell function) as a possible mechanism to explain the mortality benefit.

ELIGIBILITY:
Inclusion Criteria:

* Stage 5 Chronic Kidney Disease
* Hyperparathyroidism (PTH>300) requiring vitamin D therapy
* Age 18-80 years old
* Ability to provide informed consent

Exclusion Criteria:

* Subjects with neovascularization present, such as neoplasm, active wounds or significant retinopathy
* Subjects with contraindications or allergy to vitamin D
* Subjects currently on vitamin D therapy or a history of vitamin D therapy in the previous 60 days
* Serum phosphorus > 6
* Serum calcium > 10.5
* contraindications to nitroglycerin (such as being on sildenafil)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jula Inrig, MD, MHS, Principal Investigator — University Texas-Southwestern; Lynda Szczech, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center Dialysis Unit, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We prospectively enrolled 24 hemodialysis patients with secondary hyperparathyroidism into an open-label 30-day observational study.
Pre-assignment Details: Participants underwent review of history and meds. Hemodialysis (HD) blood was drawn. seen in vascular laboratory for testing of endothelial cell function and arterial stiffness. Doxercalciferol was initiated at dose of 2 mcg IV 3x/wk or 4 mcg IV 3x/wk. After 30 days of medication, repeat blood drawn and repeat testing in vascular laboratory.
Groups:
- Pre Doxercalciferol/Post Doxercalciferol: all end stage renal disease patients with secondary hyperparathyroidism who are vitamin D naive
  compared pre- and post doxercalciferol.
Period: Overall Study
Arm/Group | Pre Doxercalciferol/Post Doxercalciferol
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Pre-post Comparison: ESRD: all patients with secondary hyperparathyroidism who are vitamin D naive
  doxercalciferol : 2 or 4 mcg
Arm/Group | Pre-post Comparison
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Cell Function
Description: Endothelial cell function was assessed by performing flow mediated vasodilatation testing in a vascular laboratory prior to receiving doxercalciferol (either 2 mcg or 4 mcg 3 times per week at hemodialysis) and then after receiving the drug for 30 days.
Time Frame: 1 month
Population: prospective open-label 30-day observational study testing the effects of doxercalciferol on mediated vasodilation (FMD) among 20 dialysis pts with secondary hyperparathyroidism
Measure: Mean (Standard Deviation); unit: percent change in FMD
Groups:
- Pre-post Comparison: ESRD: all patients with secondary hyperparathyroidism who are vitamin D naive
  doxercalciferol
Arm/Group | Pre-post Comparison
Number analyzed (Participants) | 20
percent change in FMD | .23 (1.4)

ADVERSE EVENTS:
Groups:
- Pre and Post Doxicalciferol: ESRD: all patients with secondary hyperparathyroidism who are vitamin D naive
  doxercalciferol 2 mcg or 4 mcg three times per week for 1 month
Arm/Group | Pre and Post Doxicalciferol
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre and Post Doxicalciferol (N=20)
atypical chest pain (Cardiac disorders) | 1 (1) — hospitalized fot atypical chest pain after consent but prior to any/all study procedures.
diabetic gastroparesis (Metabolism and nutrition disorders) | 1 (1) — hospitalized for diabetic gastroparesis after study consent but prior to any/all study procedures.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre and Post Doxicalciferol (N=20)
serum phosphorus 10.4 (Metabolism and nutrition disorders) | 1 (1) — se po4 level 10.4 due to gross non compliance with phosphate binders

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No